CLINICAL TRIAL: NCT01252407
Title: Acute Effect of Transcutaneous Electrical Nerve Stimulation on the Sympathetic and Parasympathetic Systems in Individuals With Heart Failure
Brief Title: Acute Effect of Transcutaneous Electrical Nerve Stimulation in Heart Failure
Acronym: TensIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Rodrigo Della Méa Plentz, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TensIC
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2010-11

CONDITIONS: Improvement of Cardiovascular Autonomic Control; Reduction of Levels of Catecholamines
Keywords: Transcutaneous electrical nerve stimulation; Sympathetic nervous system; Parasympathetic nervous system; heart rate
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- tens (Experimental)
  Interventions: Other: transcutaneous electrical nerve stimulation

INTERVENTIONS:
Other: transcutaneous electrical nerve stimulation — Application of low frequency (10-Hz) and high frequency (100-Hz) TENS, in two different days

SUMMARY:
The purpose of this study is to determine acute effect the transctutaneous electrical nerve stimulation in sympathetic and parassympathetic system in individuals with heart failure.

DETAILED DESCRIPTION:
Heart failure (HF) is the inability of the heart to maintain adequate levels of blood supply to tissues. In recent years there has been an increased prevalence of heart failure (HF), in Brazil there are about two million people diagnosed with HF and 240,000 new cases per year. Thus, the IC constitutes the most serious problem now and in the fields of cardiology and public health. Sympathetic activity is increased and correlates with a worse prognosis and survival in these patients. Currently, the pharmacological blockade of the sympathetic system by chronic use of beta-blockers are commonly used to treat hyperactivity, but these interventions have side effects. The transcutaneous electrical nerve stimulation (TENS) has been used successfully to control pain in different clinical conditions and may be a noninvasive strategy to reduce drug and not the severity of increased sympathetic.

ELIGIBILITY:
Inclusion Criteria:

* Possess stable heart failure grade II or III according to NYHA;
* Ejection fraction <40% determined by echocardiography;
* Having no change in drug therapy one month before being included in the study;
* There have been Myocardial Infarction (AMI) three months before study entry;

Exclusion Criteria:

* Patients with grade IV heart failure according to NYHA;
* Acute respiratory;
* Unstable angina;
* Ventricular arrhythmia, unstable until three months before the start of the study;
* Pacemaker;
* Active smoking;
* Diabetes mellitus;
* And fever or infectious disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-03 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
differences in blood levels of catecholamines differences in blood levels of catecholamines differences in blood levels of catecholamines Differences in blood levels of catecholamines | one minute before and after transutaneous electrical nerve stimulation intervention (acute effect)
  For evaluation of catecholamines (epinephrine, norepinephrine and dopamine) will be held one antecubital venipuncture and collected into tubes containing ethylenediaminetetraacetic acid (EDTA).

SECONDARY OUTCOMES:
improvement of heart rate variability | one minute before and after transcutaneous electrical nerve stimulation intervention (acute effect)
  Temporal series of the tachogram, related to each selected segment were evaluated quantitatively considering the values of HR, total and normalized powers of low frequency (LF - 0.04 to 0.15 Hz) and high frequency (HF - 0.15 to 0.40 Hz) components of HRV and the sympato-vagal index (LF/HF).

CONTACTS AND LOCATIONS:
Locations (1):
- Rodrigo Della Méa Plentz, Porto Alegre, Rio Grande do Sul, Brazil